CLINICAL TRIAL: NCT05877456
Title: Validation of the Global Polypectomy Assessment Tool (GPAT) - a Novel Online Assessment Tool for Any Colorectal Polypectomy
Brief Title: Validation of the Global Polypectomy Assessment Tool (GPAT)
Acronym: GPAT
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0597
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Adenoma; Colorectal Polyp; Colo-rectal Cancer
Keywords: colonoscopy; polypectomy; quality in endoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Colorectal polypectomy is offten incompletely performed with high variability between endoscopists, resulting in interval cancer or repeated procedures. Current available scoring systems for polypectomy technique are lacking in different areas so the investigators developed the Global Polypectomy Assessment Tool (GPAT) which is an online video-based assessment tool for any colorectal polypectomy.

The goal of the study is to assess the validity of GPAT through demonstrating the inter-rater agreement (Fleiss Kappa (κ)). GPAT has 20 items, contains evidence-based statements to aid interpretation, calculates an overall quality score and a complexity score.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy worldwide and the second leading cause of cancer related death with approximately 880 792 deaths every year (9,2% of the global yearly 9.6 million cancer deaths). This is linked with a significant and increasing annual economic cost1.

Screening for polyps is mostly done by performing a colonoscopy, which is considered the golden standard for screening and removal of polyps and has been proven to reduce the global colorectal cancer burden significantly2,3. Endoscopic removal of polyps is preferred because of its efficiency, cost-effectiveness and safety in comparison to surgery4.

Incomplete polyp resection may contribute significantly to the development of so called 'interval cancers'5,6. These comprise up to 6% of newly diagnosed CRC cases and occur during the 6 - 36 month period following complete colonoscopy. Incompetent removal of polyps leads to higher recurrence rates, more hospitalizations and the use of standard surgery which has greater risks and is costlier7. Using the appropriate technique, depending on the size and aspect of the polyps, reduces recurrence-rates significantly and should therefore be pursued.

There is currently very little known about training for polypectomy. An international consensus on quality metrics of polypectomy still doesn't exist since the criteria for what makes a well-performed polypectomy have still not been identified. Many of the current endoscopists have never even received any training in polypectomy. A 3.4-fold difference in resection rates was found between gastroenterologist who knew they were being observed by using the Direct Observation of Polypectomy Skills competency score (DOPyS)8,9. This stresses the need for a standardized international training program. In countries where guidelines are available, not all endoscopy-trainers are aware of them nor do they apply them for evaluation of their trainees, even though it has been proven to augment a trainee's skills when he/she's given a report card10,11.

Attempts to develop score systems have already been made but each has its own restrictions. The DOPyS score system lacks in certain areas: it does not take the difficulty of the procedure into account and demands training of the assessor to make it reliable. The fact that a training is needed for DOPyS is a factor that's holding it back for international use. Procedure numbers and current quality indicators (including adenoma detection rate or withdrawal time) are not sufficient to account for good clinical competence12. So current tools are difficult to use, not accessible to all and are using outdated and debunked quality metrics. Therefore a new tool with new quality metrics should be easily accessible, easy to use and preferably have excellent interobserver reliability (even without training the assessor). For evaluation of polyps <1cm, which are the most frequent ones, many categories of the DOPyS were non-applicable.

With training moving away from a numbers-based competency, and current score systems lacking in different aspects, the identification of quality metrics for polypectomy and implementation of them into a new score-system, has become more and more pressing.

This led to the development of a new score system: the Global Polypectomy Assessment Tool (GPAT), by Tate et al. This score-system has been established based upon the Delphi technique13 what enforces the content-validity of this score-system. For its development, an online questionnaire was sent to 11 international experts in the field of EMR (Endoscopic Mucosal Resection). These experts were chosen because of their international recognition for performing outstanding polypectomies. The tool has 16 categories. Each category has several questions and generates a score. Depending on which questions are relevant to the polypectomy that the participants are assessing, more or less points can be gained. If the polypectomy is more difficult, the difficulty-score will rise and subsequently, there will be more points to be scored. This way the scoring system adapts to the difficulty of the polypectomy. This is important since no two polypectomies are the same and therefore different scoring-criteria are relevant depending on the polyp. This is a major difference in comparison to the DOPyS which does not adapt to the difficulty of the procedure.

Two scores are generated by this tool. The first score provides an indication on the quality of the polypectomy. The second score gives an indication on the difficulty of the polypectomy based upon the difference between the complexity of the assessed procedure and the maximum possible complexity. If some categories or questions are not relevant, it does not affect the score. The number of questions per category differs as well as the possible answers for each question. The score-system is web-based.

This scoring system was already validated using standardized videos of colorectal polypectomy and in a real-life endoscopy setting by this research group. In this study the investigators will correlate GPAT scores to key performance indicators for colonoscopy and polypectomy including caecal intubation rate, caecal photography score, withdrawal time, sedation usage, intra- and post-procedural bleeding, perforation and rate of recurrence. Through this comparison the investigators can assess whether an increase in GPAT scores correlates to a better patient outcome after polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists of varying abilities and grades
* Adult patients undergoing a polypectomy who agree to participate

Exclusion Criteria:

* Endoscopist does not consent to inclusion
* Patient does not consent to inclusion
* Patients <18 y

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopists of varying abilities and grades Adult patients undergoing a polypectomy who agree to participate
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
To validate the GPAT (global polypectomy assesment tool) scoring tool for polypectomy using key performance indicators. | up to 1 year
  Two scores are generated by this tool. The first score provides an indication on the quality of the polypectomy. This comprises of 6 domains: global competencies, injection, snare placement, safety checks, defect assessment, accessory techniques. The second score gives an indication on the difficulty of the polypectomy based upon the difference between the complexity of the assessed procedure and the maximum possible complexity (Size, morphology, site, access and 4 plus criteria: Size > 40mm, non granular morfology, non lifting polyp/previously attempted, ileocaecal valve, diverticular or appendiceal orifice involvement). If some categories or questions are not relevant, it does not affect the score. The number of questions per category differs as well as the possible answers for each question. The score-system is web-based.
  The maximum score for the first part of the tool is 105. For the indication on the difficulty of the polypectomy the maximum score is 17.

CONTACTS AND LOCATIONS:
Locations (1):
- uz Gent, Ghent, Gent, Belgium

REFERENCES:
- [Derived] Smeets S, Argenziano ME, De Crem AC, Desomer L, Anderson J, Bhandari P, Boskoski I, Bugajski M, Bourke MJ, Debels L, Heitman SJ, Kashida H, Lee RRT, Lyutakov I, Rivero-Sanchez L, Schoonjans C, Thomas-Gibson S, Thorlacius H, Fuccio L, Tham TC, Bisschops R, Tate DJ. Validation of the GPAT - the Global Polypectomy Assessment Tool: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2025 May;57(5):555-566. doi: 10.1055/a-2541-4028. Epub 2025 Mar 14. PMID 40086890